CLINICAL TRIAL: NCT06996964
Title: The Relationship Between Smartphone Use and Headache and Posture Disorders in University Students
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tuğçe Poyraz İşleyen, Lecturer, Bahçeşehir University
Other Study IDs: E-85646034-604.01-101665
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Headache; Postural; Defect
Keywords: headache; posture disorders; smartphone use
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore how smartphone use may be linked to headaches and posture problems in university students. With smartphones being a big part of daily life, many people spend long hours looking down at screens, which could affect their physical health.

DETAILED DESCRIPTION:
This cross-sectional descriptive study aims to investigate the effects of smartphone use on headaches and postural disorders in university students. Specifically, the study explores the relationship between smartphone usage habits, frequency and severity of headaches, and postural changes among individuals aged 18-25 years.

Background and Rationale:

Headaches are one of the most common neurological disorders and are considered the second leading cause of years lived with disability worldwide. The lifetime prevalence of headache is very high (approximately 96%), with a significantly higher rate in women. Among primary headache types, tension-type headache accounts for about 40% and migraine for around 10%. According to the International Classification of Headache Disorders, 3rd edition (ICHD-3), headaches are classified as primary or secondary.

As mobile and smartphone usage continues to increase globally, concerns have emerged regarding their potential health impacts. These devices emit electromagnetic fields (EMF), which may affect brain activity, blood circulation, and even DNA. Previous studies have indicated that smartphone use may be associated with health issues such as headaches, neck and shoulder pain, dizziness, stress, and sleep disturbances-especially in adolescents, where headache complaints linked to mobile phone use are seen in 10-20% of cases. However, the current literature includes conflicting evidence regarding this relationship.

One of the key postural problems associated with frequent smartphone use is Forward Head Posture (FHP), characterized by the head being positioned forward in relation to the shoulders. FHP places increased mechanical stress on the cervical spine, restricts the range of motion, and may negatively affect balance control, even in asymptomatic individuals.

This study aims to contribute to the growing body of literature by evaluating the relationship between smartphone use, headache severity, and posture health in a university student population.

Study Design:

The study is a descriptive, cross-sectional observational study.

Study Population:

The target population includes university students aged between 18 and 25 years. The sample size was calculated using the Raosoft sample size calculator. Based on a 90% confidence level and 10% margin of error for a population of 800 students from the Physiotherapy and Rehabilitation Department of Bahçeşehir University, the required minimum sample size is 63 participants.

Inclusion Criteria:

Individuals aged 18-25 years

Having experienced chronic headache symptoms for at least the past 3 months

Exclusion Criteria:

History of surgery on the cervical, thoracic, or lumbar spine

Diagnosis of rheumatoid arthritis or other musculoskeletal disorders

History of trauma within the past 6 months

Study Timeline:

The data collection will begin upon ethical approval and is expected to be completed within 6 months.

Data Collection Tools:

Demographic Information Form:

Collects participant data including age, sex, height, weight, and education level.

Smartphone Usage Questionnaire:

This form assesses daily smartphone usage duration, body posture during use, headache frequency, and associated symptoms. It also includes questions on strategies to reduce smartphone use and ergonomic habits.

Smartphone Addiction Scale - Short Form (SAS-SF):

Developed by Kwon et al., this 10-item, six-point Likert scale evaluates participants' risk of smartphone addiction. Scores range from 10 to 60, with higher scores indicating higher addiction risk. Cut-off points are 31 for males and 33 for females.

New York Posture Rating Chart:

This tool evaluates posture across 13 body segments. Each item is scored as 1 (severe deviation), 3 (moderate deviation), or 5 (normal posture), with total scores ranging from 13 to 65. Higher scores reflect better postural alignment.

Visual Analog Scale (VAS):

Used to assess the severity of headaches. Participants indicate their perceived pain intensity on a 10 cm horizontal line, where 0 = "no pain" and 10 = "worst imaginable pain." They will rate their headache intensity both during and after smartphone use.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-25 years
* Having experienced chronic headache symptoms for at least the past 3 months

Exclusion Criteria:

* History of surgery on the cervical, thoracic, or lumbar spine
* Diagnosis of rheumatoid arthritis or other musculoskeletal disorders
* History of trauma within the past 6 months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population includes university students aged between 18 and 25 years.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | day 1
  Collects participant data including age, sex, height, weight, and education level.
Smartphone Usage Questionnaire | day 1
  This form assesses daily smartphone usage duration, body posture during use, headache frequency, and associated symptoms. It also includes questions on strategies to reduce smartphone use and ergonomic habits.
Smartphone Addiction Scale - Short Form (SAS-SF) | day 1
  Developed by Kwon et al., this 10-item, six-point Likert scale evaluates participants' risk of smartphone addiction. Scores range from 10 to 60, with higher scores indicating higher addiction risk. Cut-off points are 31 for males and 33 for females.
New York Posture Rating Chart | day 1
  This tool evaluates posture across 13 body segments. Each item is scored as 1 (severe deviation), 3 (moderate deviation), or 5 (normal posture), with total scores ranging from 13 to 65. Higher scores reflect better postural alignment.
Visual Analog Scale (VAS) | day 1
  Used to assess the severity of headaches. Participants indicate their perceived pain intensity on a 10 cm horizontal line, where 0 = "no pain" and 10 = "worst imaginable pain." They will rate their headache intensity both during and after smartphone use.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğçe Poyraz Isleyen, Istanbul, Istanbul, Turkey (Türkiye)